CLINICAL TRIAL: NCT04430049
Title: Impact of the Restrictive Visiting Policy During the Covid-19 Pandemic on Anxiety, Depression and Post-traumatic Stress Disorder for Relatives of ICU Patients
Brief Title: Impact of Covid-19 Restrictive Measure on Anxiety, Depression and PTSD for Relatives of ICU Patients
Acronym: HAD-Covid
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2020 HAD-Covid
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2020-06

CONDITIONS: Covid-19; Family Members; Critical Illness
Keywords: Covid-19; Family; Anxiety; Depression; Post-traumatic stress disorder; Intensive Care Unit; Visitation
MeSH Terms: conditions — COVID-19; Critical Illness; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- no visitation group: relatives cannot visit ICU patient during Covid pandemic period in France
  Interventions: Procedure: Covid ICU containment measures
- restrictive visitation group: relatives have restriction to visit ICU patient during Covid pandemic period in France
  Interventions: Procedure: Covid ICU containment measures
- open visitation group: relatives can visit ICU patient during no Covid period in France
  Interventions: Procedure: Covid ICU containment measures

INTERVENTIONS:
Procedure: Covid ICU containment measures — The french containment measures during Covid-19 pandemic result in a restrictive visitation for relatives in ICU

SUMMARY:
To limit the pandemic Covid-19 infection, the French government imposed a closure of all Intensive Care Unit (ICU). The family's visitations are prohibited during active Covid -19 pandemic in 2020 and in 2021. This restrictive visit policy could result in an increase in symptoms of anxiety, depression or post-traumatic stress disorder for relatives of ICU patients. The aim of this study is to compare symptoms of anxiety, depression or post-traumatic stress for relatives of ICU patients during Covid period with those during no Covid period (2020 and 2021) with those no Covid period (2022)

DETAILED DESCRIPTION:
Observational multicenter study

Three groups are compared:

* no visitation group. Enrollment during the application of national containment measures to limit Covid pandemic in France: March to June 2020
* restrictive visitation group. Enrollment during the application of national containment measures to limit Covid pandemic in France: March to June 2021
* open visit group. Enrollment during a no Covid period without restrictive visitation: March to June 2022 The primary objective is to compare the Hospital Anxiety and Depression Scale (HADS) for relative at 3-6 months after the ICU patient discharge between the three groups The secondary objectives are
* to compare the Post-Traumatic Stress Disorder (PTSD) for relative at 3-6 months after the ICU patient discharge between the three groups
* to compare the prevalence of significant symptoms of both anxiety and depression for relative at 3-6 months after the ICU patient discharge between the three groups
* to compare the prevalence of significant PTSD-related symptoms for relative at 3-6 months after the ICU patient discharge between the three groups
* to identify the factor associated with significant symptoms of both anxiety and depression
* to identify the factor associated with significant PTSD-related symptoms

ELIGIBILITY:
Inclusion Criteria:

* Relative of patient who was admitted in ICU and treated with invasive mechanical ventilation administration during 24hours at least.

Exclusion Criteria:

* Relative who declines the enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relative of patient who was admitted in ICU and treated with mechanical ventilation or non-invasive ventilation or high flow oxygen or amine administration during 24hours at least.
Sampling Method: Non-Probability Sample
Enrollment: 811 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Anxiety | Between 3 and 6 months
  Anxiety for relative of ICU patient will be measured by the Hospital Anxiety and depression scale (HADS) assessed between 3 and 6 months after the ICU discharge of patient.
  HADS ranges from 0 to 42; higher scores indicate worse symptoms.
Depression | Between 3 and 6 months
  Anxiety for relative of ICU patient will be measured by the Hospital Anxiety and depression scale (HADS) assessed between 3 and 6 months after the ICU discharge of patient.
  HADS ranges from 0 to 42; higher scores indicate worse symptoms.

SECONDARY OUTCOMES:
post-traumatic stress disorder | between 3 and 6 months
  Impact of post traumatic stress disorder for relative of ICU patient will be measured with the Event scale revised (IES-R) assessed between 3 and 6 months after the ICU discharge of patient.
  IES-R ranges from 0 to 88; higher scores indicate worse symptoms

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - University hospital, Clermont-Ferrand, Clermont-Ferrand, Auvergne
  - CH Aurillac, Aurillac
  - CH Cannes, Cannes
  - Centre Jean Perrin, Clermont-Ferrand
  - CH Grenoble, Grenoble
  - CH Le Puy-en-Velay, Le Puy-en-Velay
  - University hopistal, Lyon, Lyon
  - CH Moulins, Moulins
  - CH Périgueux, Périgueux
  - CH Rodez, Rodez
  - CH Vichy, Vichy